CLINICAL TRIAL: NCT07057869
Title: Comparison of the Effects of Different Ultrasound Treatment Durations on Pain and Physical Function in Patients With Knee Osteoarthritis
Brief Title: Ultrasound Duration Effects on Knee Osteoarthritis Pain and Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: KTO Karatay University (Other)
Responsible Party: Principal Investigator, Mustafa Savaş Torlak, Associate Professor, KTO Karatay University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KaratayMST-2
Record Dates: First submitted 2025-06-30; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Knee Osteoarthristis
Keywords: Knee Osteoarthritis, Ultrasound Therapy, Pain Management, Physical Function
MeSH Terms: conditions — Osteoarthritis, Knee; Agnosia

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial where 60 patients with knee osteoarthritis are randomly assigned to three groups receiving ultrasound therapy for 5, 10, or 15 minutes respectively. All groups receive conventional treatment alongside ultrasound therapy. The effects on pain and physical function are evaluated before and after a 4-week treatment period.
Masking Description: This study is an open-label trial where both patients and treating physiotherapists are aware of the ultrasound treatment duration. Outcome assessors are blinded to group assignments to reduce assessment bias.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 5-minute Ultrasound Group (Experimental): Patients receive 5 minutes of pulsed ultrasound therapy (1 W/cm², 1 MHz) alongside conventional treatment for 4 weeks.
  Interventions: Procedure: 5-minute Ultrasound Group
- 10-minute Ultrasound Group (Experimental): Patients receive 10 minutes of pulsed ultrasound therapy (1 W/cm², 1 MHz) alongside conventional treatment for 4 weeks.
  Interventions: Procedure: 10-minute Ultrasound Group
- 15-minute Ultrasound Group (Experimental): Patients receive 15 minutes of pulsed ultrasound therapy (1 W/cm², 1 MHz) alongside conventional treatment for 4 weeks.
  Interventions: Procedure: 15-minute Ultrasound Group

INTERVENTIONS:
Procedure: 5-minute Ultrasound Group — Pulsed ultrasound therapy applied at 1 W/cm² intensity and 1 MHz frequency for 5 minutes per session, 4 weeks duration.
  Arms: 5-minute Ultrasound Group
Procedure: 10-minute Ultrasound Group — Pulsed ultrasound therapy applied at 1 W/cm² intensity and 1 MHz frequency for 10 minutes per session, 4 weeks duration.
  Arms: 10-minute Ultrasound Group
Procedure: 15-minute Ultrasound Group — Pulsed ultrasound therapy applied at 1 W/cm² intensity and 1 MHz frequency for 15 minutes per session, 4 weeks duration.
  Arms: 15-minute Ultrasound Group

SUMMARY:
This study aims to compare the effects of different ultrasound treatment durations on pain and physical function in patients with knee osteoarthritis. Sixty sedentary volunteers aged 18-85 with diagnosed knee osteoarthritis will be randomly assigned to three groups receiving ultrasound therapy for 5, 10, or 15 minutes, respectively, alongside conventional treatment. Pain and physical function will be assessed using the Visual Analog Scale (VAS), WOMAC Osteoarthritis Index, and 2-minute walk test at baseline and after 4 weeks of treatment. The results will help determine the optimal ultrasound treatment duration for improving symptoms in knee osteoarthritis patients.

DETAILED DESCRIPTION:
This clinical trial investigates the effects of different ultrasound therapy durations on pain relief and physical function improvement in patients with knee osteoarthritis. Sixty sedentary individuals aged 18 to 85 years diagnosed with knee osteoarthritis will be enrolled and randomly assigned to three groups receiving ultrasound treatment for 5, 10, or 15 minutes, respectively, alongside conventional therapy (such as hot packs, TENS, etc.).

Ultrasound therapy will be applied by a qualified physiotherapist at 1 W/cm² intensity and 1 MHz frequency in pulsed mode, for four weeks. Evaluations will be conducted at baseline and after treatment completion, using the Visual Analog Scale (VAS) for pain assessment, WOMAC Osteoarthritis Index for physical function, and a 2-minute walk test to measure walking performance.

This study aims to provide scientific evidence on the optimal ultrasound treatment duration for knee osteoarthritis, contributing to improved rehabilitation protocols. The findings will be prepared for publication in an international peer-reviewed journal.

ELIGIBILITY:
Inclusion Criteria:

Individuals aged between 18 and 85 years Diagnosed with knee osteoarthritis Recommended for ultrasound therapy as part of routine physical therapy Willing to participate voluntarily and provide written informed consent

Exclusion Criteria:

History of acute knee trauma Individuals with contraindications to ultrasound therapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-20 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Pain Intensity (VAS) | Baseline, 4 weeks
  Assessment of knee pain intensity using the Visual Analog Scale (VAS) at baseline and after 4 weeks of treatment.
Physical Function (WOMAC) | Baseline, 4 weeks
  Evaluation of physical function and stiffness using the WOMAC index at baseline and after 4 weeks of treatment.

SECONDARY OUTCOMES:
Walking Distance (2-Min Walk) | Baseline, 4 weeks
  Distance covered in 2 minutes walking test at baseline and after 4 weeks of treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- KTO Karatay Üniversitesi, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Eyigor S, Karapolat H, Ibisoglu U, Durmaz B. [Does transcutaneous electrical nerve stimulation or therapeutic ultrasound increase the effectiveness of exercise for knee osteoarthritis: a randomized controlled study]. Agri. 2008 Jan;20(1):32-40. Turkish. PMID 18338277
- [Result] Paget C, Chow MT, Duret H, Mattarollo SR, Smyth MJ. Role of gammadelta T cells in alpha-galactosylceramide-mediated immunity. J Immunol. 2012 Apr 15;188(8):3928-39. doi: 10.4049/jimmunol.1103582. Epub 2012 Mar 12. PMID 22412194
- [Result] Rutjes AW, Nuesch E, Sterchi R, Juni P. Therapeutic ultrasound for osteoarthritis of the knee or hip. Cochrane Database Syst Rev. 2010 Jan 20;(1):CD003132. doi: 10.1002/14651858.CD003132.pub2. PMID 20091539
- [Result] Huang MH, Lin YS, Lee CL, Yang RC. Use of ultrasound to increase effectiveness of isokinetic exercise for knee osteoarthritis. Arch Phys Med Rehabil. 2005 Aug;86(8):1545-51. doi: 10.1016/j.apmr.2005.02.007. PMID 16084806
- [Result] Cetin N, Aytar A, Atalay A, Akman MN. Comparing hot pack, short-wave diathermy, ultrasound, and TENS on isokinetic strength, pain, and functional status of women with osteoarthritic knees: a single-blind, randomized, controlled trial. Am J Phys Med Rehabil. 2008 Jun;87(6):443-51. doi: 10.1097/PHM.0b013e318174e467. PMID 18496246